CLINICAL TRIAL: NCT07113847
Title: Effectiveness of Resin-Based Desensitizer and Laser, Compared to Fluoride Varnish in Management of Dentine Hypersensitivity in Non-carious Cervical Lesions
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Amr Shalaby, Demonstrator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-011
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dentin Hypersensitivity, Non-carious Cervical Lesions, Bioactive Glass Air Polishing, S-PRG; Dentin Hypersensitivity; Dentin Desensitizing Agents; Desensitization
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: 84 patients who fulfill the inclusion criteria will be enrolled to the study. For every patient a tooth of complain which fulfill the inclusion criteria will be selected, so the total number of included teeth will be 84 teeth. Teeth will be classified into 4 groups according to the type of desensitizer used. Where in group 1 (G1) patients will be randomly assigned to "Resin-Based Desensitizer", in group 2 (G2) patients will be randomly assigned to "Laser Desensitizer", in group 3 (G3) patients will be randomly assigned to "Combination of Laser + Resin-Based Desensitizer", and in group 4 (G4) patients will be randomly assigned to "Fluoride-Based Desensitizer". For every patient, sensitivity test will be done using visual analogue scale immediately after application, three months after application and six months after application. Table 1 shows the variables of the study,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resin-Based Desensitizer (Active Comparator)
  Interventions: Biological: Resin-Based Desensitizer
- Laser Desensitizer (Active Comparator)
  Interventions: Device: Laser Desensitizer
- Combination of Laser + Resin-Based Desensitizer (Active Comparator)
  Interventions: Biological: Resin-Based Desensitizer; Device: Laser Desensitizer
- Fluoride-Based Desensitizer (Active Comparator)
  Interventions: Biological: Fluoride-Based Desensitizer

INTERVENTIONS:
Biological: Resin-Based Desensitizer — resin desensitizing agent
  Arms: Combination of Laser + Resin-Based Desensitizer; Resin-Based Desensitizer
Device: Laser Desensitizer — Low-power Diode laser
  Arms: Combination of Laser + Resin-Based Desensitizer; Laser Desensitizer
Biological: Fluoride-Based Desensitizer — Fluoride-based varnish
  Arms: Fluoride-Based Desensitizer

SUMMARY:
84 patients who fulfill the inclusion criteria will be enrolled to the study. For every patient a tooth of complain which fulfill the inclusion criteria will be selected, so the total number of included teeth will be 84 teeth. Teeth will be classified into 4 groups according to the type of desensitizer used. Where in group 1 (G1) patients will be randomly assigned to "Resin-Based Desensitizer", in group 2 (G2) patients will be randomly assigned to "Laser Desensitizer", in group 3 (G3) patients will be randomly assigned to "Combination of Laser + Resin-Based Desensitizer", and in group 4 (G4) patients will be randomly assigned to "Fluoride-Based Desensitizer". For every patient, sensitivity test will be done using visual analogue scale immediately after application, three months after application and six months after application. Table 1 shows the variables of the study, and Table 2 shows the variables of the study.

Each patient's name will be replaced with a case number within the group to protect the privacy of medical information and data of the patients.

DETAILED DESCRIPTION:
1. Participants Randomization and Allocation:

   Using computer generated randomization, the participants will be allocated randomly into four equal groups.

   The sequentially numbers that will be generated, will be placed in opaque envelope until the intervention and each participant will be asked to select an envelope that determine which group of intervention he will be assigned.
2. Interventions:

   Grouping 84 patients who fulfill the inclusion criteria will be enrolled to the study. For every patient a tooth of complain which fulfill the inclusion criteria will be selected, so the total number of included teeth will be 84 teeth. Teeth will be classified into 4 groups according to the type of desensitizer used. Where in group 1 (G1) patients will be randomly assigned to "Resin-Based Desensitizer", in group 2 (G2) patients will be randomly assigned to "Laser Desensitizer", in group 3 (G3) patients will be randomly assigned to "Combination of Laser + Resin-Based Desensitizer", and in group 4 (G4) patients will be randomly assigned to "Fluoride-Based Desensitizer". For every patient, sensitivity test will be done using visual analogue scale immediately after application, three months after application and six months after application. Table 1 shows the variables of the study, and Table 2 shows the variables of the study.

   Each patient's name will be replaced with a case number within the group to protect the privacy of medical information and data of the patients.

   Clinical Procedures:

   Controlled air stimulus (Evaporative) will be applied on the tooth of complain, using dental syringe adjusted 40-65 psi directed perpendicular at a distance 1-3 mm from the exposed dentine. The patient should point out the degree of sensitivity on the VAS scale (0-10) chart the degree of pain. (VAS >5). Plastic card with figures of facial expressions expressing degree of pain, color coded, and numbers guided was used to ease the process of figuring out the degree of pain.

   For Resin-Based Desensitizer Group Cheek retractors and high-volume suction will be used for keeping dry and visible field as much as possible. The teeth will be thoroughly cleaned, and the surfaces will be air-dried. After proper dryness and with the aid of a micro-brush, resin-based desensitizer will be applied to the sensitive areas. Application time, and technique will be done according to manufacturer instructions. Then it will be cured using LED curing unit according to manufacturer instructions.

   For Laser Group The teeth will be thoroughly cleaned, and the surfaces will be air-dried. Low-power Diode laser will be used with the recommended parameters of the manufacturer for dentine hypersensitivity. The tip will be placed perpendicular to the tooth surface and moved over the lesion for the specified direction and time.

   For Combination Group Laser will be applied in the same parameters and technique as for the laser group, then it will be followed by the application of resin-based desensitizer following same instructions as the resin-based desensitizer group.

   For Fluoride-Based Group (Comparator) The teeth will be thoroughly cleaned, and the surfaces will be air-dried. The Fluoride-based varnish will be applied to the tooth structure using a micro-brush. Number and technique of application will be done according to manufacturer instructions.

   Post-Operative Instructions All patients will be instructed to avoid eating and drinking for an hour, avoid brushing or flossing for at least 4-6 hours.
3. Outcomes:

Assessment of Outcome The post-operative hypersensitivity assessment will be performed for immediately, three months and six months after application using visual analogue scale (VAS).[19] It is a horizontal line graded from 1 to 10 with a descriptor at its far-left end indicating no pain, and at its far-right end indicating the worst possible pain. Illustration of facial expressions with color codes was added below the 10-centimeter line Visual Analog Scale.[20] (Figure 1). Assessment of the final outcome

ELIGIBILITY:
Inclusion Criteria of Participants:

1. Males or Females
2. 18 -50 years.
3. Not received antibiotic therapy for 1 month before sampling.
4. Good oral hygiene.
5. Co-operative patients approving the trial.
6. Compliant patients.

Exclusion Criteria of Participants:

1. Pregnancy.
2. Systemic disease or severe medical complications.
3. Patients who did any periodontal surgeries within the previous 6 months.
4. Patients with bad oral hygiene.
5. Patients who are allergic to any ingredients used in the study.
6. Xerostomia.
7. Lack of compliance.

Inclusion Criteria of Teeth:

1. Non carious lesions.
2. Cervical lesions.
3. Teeth with DH, VAS >5.

Exclusion Criteria of Teeth:

1. Carious teeth.
2. Chipped teeth.
3. Teeth with mobility Grade 2 or 3.
4. Teeth with probing depth more than 4 mm.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | 0,3,6 months
  post-operative hypersensitivity assessment with the visual analogue scale from 0-10 with 0 is the minimum sensitivity record and 10 is the maximum sensitivity record

CONTACTS AND LOCATIONS:
Locations (1):
- BUE, Cairo, El Shorouk City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All Data are available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year